CLINICAL TRIAL: NCT00473278
Title: Analysis of Human Tear Proteins in Children: A Pilot Study to Describe the Tear Film Proteome of Pediatric Patients Undergoing Ophthalmic Examination.
Brief Title: Analysis of Human Tear Proteins in Children
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 06-1067
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Eye Disease
Keywords: tear protein
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The significance of our study is in the importance of understanding the quality and quantity of proteins in the human tear film, and any unique aspects of tears in children. This pilot study will provide data to plan prospective research to better delineate the utility of tear proteins in diagnosing and following disease status in a non-invasive fashion.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age
* A parent or legal guardian provide written informed consent to participate
* Able to cooperate with tear sample collection, or a previously planned sedation for other medical purposes

Exclusion Criteria:

* Age greater than or equal to 18 years
* Patients' parents or legal guardians who refuse to sign study consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children less than 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Proteome of Human Tears | Single Exam

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — Rocky Mountain Lions Eye Institute
Locations (1):
- The Childrens Hospital, Denver, Colorado, United States